CLINICAL TRIAL: NCT01558375
Title: A Double-blind, Randomized, Placebo-controlled Clinical Trial of the Safety and Efficacy of Anakinra in Patients With Hidradenitis Suppurativa
Brief Title: Anakinra in Hidradenitis Suppurativa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Evangelos J. Giamarellos-Bourboulis, M.D., Associate Professor of Medicine, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HIDRA03
Record Dates: First submitted 2012-03-15; First posted 2012-03-20 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Water; Injections; Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Water for injection (Placebo Comparator): Placebo syringes will contain 0.67ml of sterile water for injection. This will be injected daily for 12 weeks.
  Interventions: Drug: Water for injection
- Anakinra (Experimental): Anakinra will be supplied in single use pre-filed glass syringes with 27-gauge needles. Anakinra syringe will contain 100mg of anakinra at a volume of 0.67 ml. This will be injected subcutaneously daily for 12 weeks.
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Water for injection — Placebo syringes will contain 0.67ml of sterile water for injection. This will be injecteda daily for 12 weeks.
  Other Names: Sterile water
  Arms: Water for injection
Drug: Anakinra — Anakinra will be supplied in single use pre-filed glass syringes with 27-gauge needles. Anakinra syringe will contain 100mg of anakinra at a volume of 0.67 ml. This will be injected subcutaneously daily for 12 weeks.
  Other Names: Recombinant human IL-1 receptor antagonist
  Arms: Anakinra

SUMMARY:
Aim of this double-blind, randomized, controlled clinical trial is to compare the safety and the efficacy of anakinra over placebo for the management of patients with hidradenitis suppurativa (HS) of Hurley II and Hurley III disease stage. Patients will be evaluated on subsequent follow-up visits. Two scores will be applied: disease activity as assessed in the protocol by the investigator; and Sartorius score. Primary efficacy endpoint will be the comparisons of visual analogue scores, of disease activity, of Sartorius score and of dermatology life quality index between the two groups of treatment over follow-up.

DETAILED DESCRIPTION:
Hidradenitis suppurativa (HS) is a chronic devastating skin disorder affecting areas rich in apocrine glands. Nodules appear in the affected areas; they progressively become swollen and rupture with the release of pus. This process occurs repeatedly leading to sinus tract formation and scars. This disease course creates a frustrating situation for the patients but also for physicians. Traditional treatments comprise short-courses of antibiotics and surgical excision. However, relapse is the rule so that HS leads to severe impairment of the quality of life. The Dermatology Quality Life Index (DQLI) for HS is 8.9 being higher than any other skin disorder.

This devastating disorder has often been neglected and considered a rare situation. However, HS seems to indiscriminately affect the global population. Although the exact epidemiology is largely unknown, the point-prevalence is reported to range between 1% and 4%. A recent large epidemiological survey in France reports 0.97% disease prevalence.

The exact pathophysiology of HS is unknown. Smoking, dietary habits and genetic predisposition have all been linked with HS. However, a recent survey by our group in 56 patients, disclosed a severe derangement of the monocyte function and of subsequent antigen processing in these patients. The percentage of natural killer (NK) cells was increased and that of CD4-lymphocytes decreased compared to healthy controls probably implying the existence of an autoimmune predilection for the disorder. We have previously demonstrated defective lipopolysaccharide (LPS)-induced production of the pro-inflammatory cytokines, tumour necrosis factor(TNF) and interleukin (IL)-6 by blood monocytes of patients with HS.

As a consequence, a hypothesis for the implication of some autoimmune of autoinflammatory mechanism in the pathogenesis of HS was started to be created over the last years. The hypothesis is further reinforced by positive results from the administration of TNF antagonists in prospective studies with limited number of patients one of these was conducted by our study group. Subcutaneous treatment with 50mg etanercept once weekly for 12 weeks in 10 patients, reduced patients' suffering, attenuated local signs of inflammation and retarded disease relapse.

Anakinra is a recombinant interleukin-1 (IL-1) receptor antagonist (IL-1Ra). Anakinra blocks the biologic activity of naturally occurring IL-1, including inflammation and cartilage degradation associated with rheumatoid arthritis, by competitively inhibiting the binding of IL-1 to the interleukin-1 type receptor, which is expressed in many tissues and organs. IL-1 is produced in response to inflammatory stimuli and mediates various physiologic responses, including inflammatory and immunologic reactions. The biological properties of anakinra and the existing clinical and laboratory data favoring a derangement of the immune response in HS, prompted to investigate whether anakinra would be efficient in the management of patients with HS.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent provided by the patient;
* age above 18 years;
* diagnosis of hidradenitis suppurativa; and
* disease of Hurley II or III severity stage

Exclusion Criteria:

* history of systemic lupus erythematosus, of rheumatoid arthritis of of seronegative inflammatory arthritis;
* any prior administration of any type of anti-TNF therapy over the last six months;
* administration of any live (attenuated) vaccine over the last 4 weeks;
* history of recurrent vein thrombosis or embolism compatible with anti-cardiolipin syndrome;
* any present or smoldering infection;
* hepatic dysfunction defined as any value of transaminases, of γ-glutamyl transpeptidase or of bilirubin> 2 x upper normal limit;
* history of haematological or solid tumor malignancy, arterial hypertension, liver cirrhosis, HIV infection, and hepatitis virus B or C infection
* history of episodes mimicking demyelinating disorders or a definite diagnosis of multiple sclerosis
* any creatinine value above 1.5 mg/dl
* intake of corticosteroids defined as daily intake of prednisone or equivalent more than 1mg/kg for the last three weeks;
* neutropenia defined as <1000 neutrophils/mm3; and
* pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The efficacy of anakinra in patients with HS of Hurley II and III stage disease. | 24 weeks
  This will be defined by the changes of scoring parameters between the two study groups over visits.

SECONDARY OUTCOMES:
The effect of anakinra in the ex vivo function of monocytes of patients with HS. | 24 weeks
  This will be defined by the differences of cytokines produced by PBMCs between the two study groups over visits.
The effect of anakinra on the time to new exacerbation | 24 weeks
  This will be defined by the differences between the two study groups over visits.
The safety of anakinra in patients with hidradenitis suppurativa | 24 weeks
  This will be assessed by the development of serious and non-serious drug-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos J Giamarellos-Bourboulis, MD, PhD, Study Chair — University of Athens, Medical School, Greece; Dimitrios Rigopoulos, MD, PhD, Principal Investigator — University of Athens, Medical School, Greece
Locations (2):
- Greece (2):
  - 2nd Department of Dermatology, ATTIKON University Hospital, Athens
  - 4th Department of Internal Medicine, ATTIKON University Hospital, Athens

REFERENCES:
- [Background] Giamarellos-Bourboulis EJ, Pelekanou E, Antonopoulou A, Petropoulou H, Baziaka F, Karagianni V, Stavrianeas N, Giamarellou H. An open-label phase II study of the safety and efficacy of etanercept for the therapy of hidradenitis suppurativa. Br J Dermatol. 2008 Mar;158(3):567-72. doi: 10.1111/j.1365-2133.2007.08372.x. Epub 2007 Dec 11. PMID 18076705
- [Background] Giamarellos-Bourboulis EJ, Antonopoulou A, Petropoulou C, Mouktaroudi M, Spyridaki E, Baziaka F, Pelekanou A, Giamarellou H, Stavrianeas NG. Altered innate and adaptive immune responses in patients with hidradenitis suppurativa. Br J Dermatol. 2007 Jan;156(1):51-6. doi: 10.1111/j.1365-2133.2006.07556.x. PMID 17199566
- [Background] Kurzen H, Kurokawa I, Jemec GB, Emtestam L, Sellheyer K, Giamarellos-Bourboulis EJ, Nagy I, Bechara FG, Sartorius K, Lapins J, Krahl D, Altmeyer P, Revuz J, Zouboulis CC. What causes hidradenitis suppurativa? Exp Dermatol. 2008 May;17(5):455-6; discussion 457-72. doi: 10.1111/j.1600-0625.2008.00712_1.x. PMID 18400064
- [Background] Pelekanou A, Kanni T, Savva A, Mouktaroudi M, Raftogiannis M, Kotsaki A, Giamarellos-Bourboulis EJ. Long-term efficacy of etanercept in hidradenitis suppurativa: results from an open-label phase II prospective trial. Exp Dermatol. 2010 Jun;19(6):538-40. doi: 10.1111/j.1600-0625.2009.00967.x. Epub 2009 Sep 16. PMID 19758320
- [Derived] Tzanetakou V, Kanni T, Giatrakou S, Katoulis A, Papadavid E, Netea MG, Dinarello CA, van der Meer JWM, Rigopoulos D, Giamarellos-Bourboulis EJ. Safety and Efficacy of Anakinra in Severe Hidradenitis Suppurativa: A Randomized Clinical Trial. JAMA Dermatol. 2016 Jan;152(1):52-59. doi: 10.1001/jamadermatol.2015.3903. PMID 26579854
- See also: Hidradenitis suppurativa foundation — http://www.hs-foundation.org